CLINICAL TRIAL: NCT00622440
Title: Phase II Study for Treatment of Anal HSIL Through Use of a Chinese Herbal Topical Cream
Brief Title: Treatment of Anal High-grade Squamous Intraepithelial Lesions (HSIL) Through Use of a Chinese Herbal Topical Cream
Acronym: AIJP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Spring Wind Herbs (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 07501; P-07-020 (Other Grant/Funding Number: Cancer Treatment Research Foundation (CTRF)); NCI-2011-03238 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2008-02-13; First posted 2008-02-25 (Estimated); Results first posted 2014-08-12 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Anus Neoplasms
Keywords: HSIL; HGAIN; AIN; neoplasia; dysplasia; TCM; Traditional Chinese Medicine
MeSH Terms: conditions — Anus Neoplasms; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: AIJP (Arnebia Indigo Jade Pearl)
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AIJP (Arnebia Indigo Jade Pearl) — Participants will administer their own treatment using 1/4 teaspoon of the cream twice daily for 48 weeks.
  Arms: 1
Drug: Placebo — Placebo twice daily for 48 weeks.
  Arms: 2

SUMMARY:
The purpose of this study is to find out if a Chinese herbal cream is effective in treating HSIL (high-grade squamous intraepithelial lesions, also known as HGAIN, or high-grade anal intraepithelial neoplasia).

DETAILED DESCRIPTION:
The purpose of this study is to test a new noninvasive topical cream, AIJP (Arnebia Indigo Jade Pearl), for treatment of precancerous anal lesions in order to prevent their progression to anal cancer. AIJP is a topical Chinese herbal cream that has been specifically designed to treat people with the cancer precursor lesions caused by human papillomavirus (HPV). In general, HPV infection is a key factor in development of cervical, anal and vulvar cancers. People with HIV are especially vulnerable to develop anal cancer associated with HPV. It is known that prior to development of anal cancer a person develops a precancerous condition known as a high-grade squamous intraepithelial lesion (HSIL). Treatment of the HSIL can prevent progression to anal cancer. Current therapies for HSIL and anal cancer are highly invasive. A new effective noninvasive topical therapy for precancerous HSIL could have a high impact on prevention of anal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Anal HSIL confirmed by biopsy no more than 30 days prior to entry
* Anal HSIL deemed not amenable to therapy or participant declines routine ablative therapy
* HIV positive
* Stable HIV treatment regimen for at least 8 weeks prior to entry
* At least 18 years of age
* Women of childbearing potential must use contraception
* Platelet count above 70,000/mm3 within 30 days prior to entry
* ANC greater or equal to 1000/mm3 within 30 days prior to entry
* Creatinine less then or equal to 1.5 times ULN within 30 days prior to entry
* AST and ALT less than or equal to 3 times ULN within 30 days prior to entry

Exclusion Criteria:

* Prior history of invasive anal, cervical, vaginal, or vulvar cancer
* Pregnancy or lactation and breast-feeding
* Must not participate in a conception process including sperm donation
* Medical or psychiatric illness that precludes ability to give informed consent or is likely to interfere with ability to comply with protocol
* Known allergy to any topical cream components
* Patients with lesions clinically suspicious per HRA examiner for early progression (less than one year) to anal cancer

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-05-14 (Actual); Primary Completion 2012-12-12 (Actual); Study Completion 2012-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Misha R Cohen, OMD, LAc, Principal Investigator — Chicken Soup Chinese Medicine; Naomi Jay, PhD, FNP, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: General information about HPV, dysplasia, and anal cancer. The website also includes a list of providers of high-resolution anoscopy (HRA). — http://www.ucsfhealth.org/adult/medical_services/cancer/cr/conditions/anal/signs.html

RESULTS

PARTICIPANT FLOW:
Groups:
- AIJP: AIJP (Arnebia Indigo Jade Pearl): Participants administer 1/4 teaspoon of AIJP cream twice daily for 48 weeks.
- Placebo: Placebo: Participants administer 1/4 teaspoon of placebo cream twice daily for 48 weeks.
Period: Baseline - Week 12 (Treatment)
Arm/Group | AIJP | Placebo
Started | 35 | 35
Completed | 31 | 34
Not Completed | 4 | 1
Not completed — Received cream but did not return | 4 | 1
Period: Week 12 - Week 48 (Treatment)
Arm/Group | AIJP | Placebo
Started | 31 | 34
Completed | 28 | 28
Not Completed | 3 | 6
Not completed — Lost to Follow-up | 3 | 5
Not completed — Not evaluable - censored from dataset | 0 | 1
Period: Week 60 (Post-treatment Follow-up Visit)
Arm/Group | AIJP | Placebo
Started | 28 | 28
Completed | 28 | 27
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AIJP | Placebo | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Customized [Number; unit: participants]
  24-39 years | 5 | 10 | 15
  40-59 years | 25 | 22 | 47
  60-74 years | 5 | 3 | 8
Sex/Gender, Customized [Number; unit: participants]
  Men | 34 | 33 | 67
  Women | 1 | 1 | 2
  MTF (transgender) | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 9
  Not Hispanic or Latino | 29 | 32 | 61
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 1 | 4 | 5
  White | 32 | 24 | 56
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Final Response of Anal High-grade Squamous Intraepithelial Lesions (HSIL)
Description: Response assessed 12 weeks after treatment.
  Late Clinical Response (LCR): HSIL present at week 48 but none at week 60, with two independent reviews in agreement that HSIL absent at week 60.
  Complete response (CR): No HSIL on histology or cytology at weeks 48 or 60 (caveat: if HSIL at week 60, blinded chart notes and photographs were reviewed by two clinicians, and decision was reached by agreement or consensus whether HSIL had been missed at week 48. Cases that reviewers independently agreed had not been missed at week 48 were considered true recurrences)
  Partial Clinical Response (PCR): HSIL on cytology with no HSIL histology, or improvement >50% in the number of lesions with HSIL, or an improvement >50% in lesion size, area, or clinical characteristics (e.g. acetowhite staining, Lugol's staining, or vascular changes were improved)
  No Response (NR): HSIL present at weeks 48 & 60 on histology, or improvement ≤ 50% in number, size, area or characteristics.
Time Frame: Baseline, Week 48, and Week 60; up to 60 weeks
Measure: Number; unit: participants
Arm/Group | AIJP | Placebo
Number analyzed (Participants) | 28 | 28
participants
  LCR | 3 | 0
  CR | 7 | 3
  PCR | 5 | 6
  NR | 13 | 19
Statistical Analysis 1: Comparison: AIJP vs Placebo; Estimated Effect Size for Phase 3 Trial; Test type: Other; p = .042, Wilcoxon rank sum; Wilcoxon Rank Sum Effect Size = 0.275 — The wilcoxon rank sum effect size ranges in strength of effect from small (0.10 - < 0.30), to medium (0.30 - < 0.50), to large (>=0.50) with a total range of 0 to 1

2. Secondary Outcome: Treatment Adherence
Description: Percent of recommended applications of cream reported in participant diary.
  >75% = Excellent >50%-75% = Good >25%-50% = Poor <25% = Non-adherent
Time Frame: Up to 48 weeks
Population: Excludes 7 AIJP participants and 6 Placebo participants who dropped out before week 48. Excludes 1 Placebo participant deemed non-evaluable.
Measure: Number; unit: participants
Arm/Group | AIJP | Placebo
Number analyzed (Participants) | 28 | 28
participants
  Excellent | 17 | 15
  Good | 9 | 6
  Poor | 1 | 4
  Non-adherent | 1 | 3

3. Secondary Outcome: Response With >50% Adherence
Description: Response assessed 12 weeks after treatment (week 60), by treatment adherence assessed at 48 weeks.
  Late Clinical Response (LCR): HSIL present at week 48 but none at week 60; two independent reviews agree HSIL absent at week 60.
  Complete response (CR): No HSIL on histology or cytology at weeks 48 or 60 (caveat: if HSIL at week 60, blinded chart notes and photographs reviewed by two clinicians, with decision by agreement or consensus whether HSIL had been missed at week 48. Cases that reviewers independently agreed had not been missed at week 48 were considered true recurrences)
  Partial Clinical Response (PCR): HSIL on cytology with no HSIL histology, or improvement >50% in number of lesions with HSIL, or improvement >50% in lesion size, area, or clinical characteristics (e.g. acetowhite staining, Lugol's staining, or vascular changes improved)
  No Response (NR): HSIL present on histology, or improvement ≤ 50% in number, size, area or characteristics.
Time Frame: Baseline, Week 48, and Week 60; up to 60 weeks
Population: Evaluable participants who finished 48 weeks of treatment and reported >50% adherence to treatment
Measure: Number; unit: participants
Arm/Group | AIJP | Placebo
Number analyzed (Participants) | 26 | 21
participants
  LCR | 3 | 0
  CR | 7 | 3
  PCR | 4 | 5
  NR | 12 | 13

4. Secondary Outcome: Response With >75% Adherence
Description: Response assessed 12 weeks after treatment (week 60), by treatment adherence assessed at 48 weeks.
  Late Clinical Response (LCR): HSIL present at week 48 but none at week 60; two independent reviews agree that HSIL absent at week 60.
  Complete response (CR): No HSIL on histology or cytology (caveat: if HSIL at week 60, blinded chart notes and photographs were reviewed by two clinicians, and decision was reached by agreement or consensus whether HSIL had been missed at week 48. Cases that reviewers independently agreed had not been missed at week 48 were considered true recurrences)
  Partial Clinical Response (PCR): HSIL on cytology with no HSIL histology, or improvement >50% in the number of lesions with HSIL, or an improvement >50% in lesion size, area, or clinical characteristics (e.g. acetowhite staining, Lugol's staining, or vascular changes were improved)
  No Response (NR): HSIL present on histology, or improvement ≤ 50% in number, size, area or characteristics.
Time Frame: Baseline, Week 48, and Week 60; up to 60 weeks
Population: Evaluable participants who finished 48 weeks of treatement and reported >75% adherence to treatment
Measure: Number; unit: participants
Arm/Group | AIJP | Placebo
Number analyzed (Participants) | 17 | 15
participants
  LCR | 3 | 0
  CR | 5 | 1
  PCR | 2 | 5
  NR | 7 | 9

ADVERSE EVENTS:
Time Frame: 60 Weeks
Arm/Group | AIJP | Placebo
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 1/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIJP (N=35) | Placebo (N=35)
Perianal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 — Superficially invasive cancer possibly present at baseline; participant non-evaluable for study outcomes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes